CLINICAL TRIAL: NCT05963321
Title: Cortical Excitability Modulation With Cerebellar Transcranial Direct Current Stimulation in Fibromyalgia: a Randomized Clinical Trial
Brief Title: Cortical Excitability Modulation With ctDCS in Fibromyalgia.
Acronym: ctDCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-0504
Record Dates: First submitted 2023-06-26; First posted 2023-07-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Fibromyalgia; Cerebellum; Transcranial direct current magnetic stimulation; Transcranial magnetic stimulation
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active cerebellum electrode and active M1 electrode (Active Comparator): * The patient will receive active cerebellar stimulation with the anode electrode positioned in the cerebellum and active cortical stimulation with the anode electrode placed in the primary motor cortex.
  * In both cerebellar and cortical stimulations, the cathode will be positioned in the contralateral supraorbital region.
  * The equipment will apply a current of 2 mA for 20 minutes.
  Interventions: Device: TDCS
- Sham cerebellar electrode and active M1 electrode (Active Comparator): * The patient will receive sham cerebellar stimulation with the anode electrode positioned in the cerebellum and active cortical stimulation with the anode electrode placed in the primary motor cortex.
  * In both cerebellar and cortical stimulations, the cathode will be positioned in the contralateral supraorbital region.
  * The equipment will apply a current of 2 mA for 20 minutes.
  Interventions: Device: TDCS
- Active cerebellum electrode and sham M1 electrode (Active Comparator): * The patient will receive active cerebellar stimulation with the anode electrode positioned in the cerebellum and sham cortical stimulation with the anode electrode placed in the primary motor cortex.
  * In both cerebellar and cortical stimulations, the cathode will be positioned in the contralateral supraorbital region.
  * The equipment will apply a current of 2 mA for 20 minutes.
  Interventions: Device: TDCS
- Sham cerebellar electrode and sham M1 electrode (Sham Comparator): * The patient will receive sham cerebellar stimulation with the anode electrode positioned in the cerebellum and sham cortical stimulation with the anode electrode placed in the primary motor cortex.
  * In both cerebellar and cortical stimulations, the cathode will be positioned in the contralateral supraorbital region.
  * The equipment will apply a current of 2 mA for 20 minutes.
  Interventions: Device: TDCS

INTERVENTIONS:
Device: TDCS — Two tDCS devices will be used simultaneously. The intervention consists of a tDCS session in which the active electrode will be located in the cerebellum and/or in the primary motor cortex (4 stimulation protocols that will be implemented; active cerebellum electrode and active M1 electrode, sham cerebellum electrode and active M1 electrode, active cerebellum and sham M1 electrode, sham cerebellar electrode and sham M1 electrode) and the cathode in the contralateral supraorbital region.

SUMMARY:
Fibromyalgia is a syndrome characterized by chronic generalized musculoskeletal pain, accompanied by other symptoms such as fatigue, sleep disturbance and depression. Complaints of memory deficit, cognitive dysfunction, headache and gastrointestinal disorders are also common. Although it is a relatively common syndrome, exist a limited effectiveness of the pharmacologycal treatment. However, In the last years new therapeutic and diagnostic options have been sought. This scenario includes the use of different techniques of non-invasive brain stimulation, such as transcranial direct current magnetic stimulation (tDCS) and transcranial magnetic stimulation (TMS), which have already had promising results in reducing pain. Based on the above, the objective of this research is to evaluate the effect of cerebellar tDCS on clinical measures of pain and cortical excitability in patients with fibromyalgia. In this study, the intervention consists of a single tDCS session in which two devices will be used simultaneously. The active electrode will be placed in the cerebellum and/or in the primary motor cortex and the cathode in the contralateral supraorbital region. It is expected that the application of this protocol will be able to have a modulatory effect on clinical pain measures. In addition to producing changes in cortical excitability as a reflection of the integration between the cerebellum-thalamus-cortical pathways.

DETAILED DESCRIPTION:
The prevalence of fibromyalgia is approximately 2.7%, with a female-to-male ratio of 3:1. Although it is a relatively common syndrome, there are many doubts regarding its diagnosis and pathophysiology. In addition to the previously mentioned questions, this pathology has high social costs due to its association with the loss of labor productivity and it is characterized by being unresponsive to pharmacological treatment. Given the limited effectiveness of available therapeutic options, new therapeutic and diagnostic options have been sought. This scenario includes the use of different techniques of non-invasive brain stimulation, such as transcranial direct current magnetic stimulation (tDCS) and transcranial magnetic stimulation (TMS), which have already had promising results in reducing pain. In addition, TMS also allows measuring parameters that help to understand the reorganization of physiological processes. In this study, TMS is used to understand the pathophysiology of fibromyalgia, while tDCS allows modulating the excitability of the neuronal membrane potential of cortical and subcortical neural networks, producing a neuromodulatory effect of the top-down type. According to the evidence, the greatest impact on pain is associated with stimulation of the primary motor cortex (M1), but recent studies have shown the possible relationship between stimulation of extracerebral regions such as the cerebellum, with an analgesic effect present in healthy individuals and patients with different pathologies. In the same way, the cortical excitability measures obtained through TMS allow us to identify the imbalance between inhibitory and excitatory systems, related to pain perception and the analgesic response of endogenous mechanisms. In this research, our objective is to evaluate the effect of cerebellar tDCS on clinical measures of pain and cortical excitability in patients with fibromyalgia. This is a randomized, double-blind, controlled clinical trial, parallel, which has as its primary outcome, the evaluation of the variations in motor evoked potential (MEP) (neurophysiological outcome) and the numerical pain scale (NPS) as a clinical outcome. Secondary outcomes include the silent period (CSP), intra-cortical facilitation (ICF) and intra-cortical inhibition (ICI) obtained through TMS, the function of the descending modulatory path of pain by the conditioned modulation test (CPM test), the Brief Pain Inventory (BPI) and the pain thresholds by heat, pressure and cold. The intervention consists of a single tDCS session in which two devices will be used simultaneously. The active electrode will be placed in the cerebellum and/or in the primary motor cortex (4 stimulation protocols that will be implemented; active cerebellum electrode - active M1 electrode, sham cerebellum electrode - active M1 electrode, active cerebellum-M1 sham electrode, sham cerebellum electrode-M1 sham electrode) and the cathode in the contralateral supraorbital region. The equipment will apply a current of 2 mA for 20 minutes. In total, there will be 92 patients, divided into 4 intervention blocks and composed of 23 individuals each.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed women aged 18 to 65 years; who can read and write
* Confirmed diagnosis of fibromyalgia according to the criteria of the American College of Rheumatology (2010-2016).
* Pain score equal to or greater than 4 on the Numerical Pain Scale (Score 0-10) on most days in the last 3 months.

Exclusion Criteria:

* Reside outside Porto Alegre area.
* Confirmed pregnancy
* Contraindications to TMS and tDCS: metallic implant in the brain; medical devices implanted in the brain, heart pacemaker; cochlear implant; history of alcohol or drug abuse in the last 6 months; neurological pathologies; hx of head trauma or neurosurgery; decompensated systemic diseases and chronic inflammatory diseases (lupus, rheumatoid arthritis, Reiter's syndrome); uncompensated hypothyroidism; personal history of cancer, past or undergoing treatment.
* Participants with diagnosis or recent contact with COVID will be excluded.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in motor evoked potential (MEP). | Up to 60 minutes after tDCS onset.
  Change from before and after tDCS onset on MEP. Assessed by a variation in the amplitude obtained by 20 stimuli with an intensity of 120% of the MT. The MEP will be considered the arithmetic mean of the amplitude of the wave recorded by the EMG.
Change in pain level | Up to 60 minutes after tDCS onset.
  The study assessed the change in pain scores before and after tDCS onset using the Numerical Pain Scale (NPS). The NPS scores range from zero (no pain) to a maximum of ten (severe pain).

SECONDARY OUTCOMES:
Change in the Brief Pain Inventory (BPI) score | Up to 15 days after tDCS onset.
  It is a quick, simple, and easy-to-apply questionnaire that allows a multidimensional pain assessment to be carried out. The BPI consists of 15 items that determine the severity, existence, location, functional interference, applied therapeutic strategies, and efficacy of pain treatment. In the research, this questionnaire will be implemented at baseline, 8 and 15 days after tDCS onset.
Change in Function of corticospinal pathway | Up to 60 minutes after tDCS onset.
  Measures of cortical excitability obtained through TMS include the silent period (CSP),intra-cortical facilitation (ICF) and intra-cortical inhibition (SICI). The TMS measures will be performed at two different times: before and after tDCS onset.
change in conditioned pain modulation (CPM) | Up to 60 minutes after tDCS onset.
  Conditioned pain modulation (CPM) is an experimental psychophysical measure that assesses supraspinal descending inhibitory mechanisms of pain modulation. In practice, a constant noxious stimulus (conditioning stimulus) is applied to one part of the body and a phasic stimulus (stimulus to be tested) to a distant part of the body before, during, and after the conditioning stimulus. The CPM is analyzed through the reduction that occurs in the perception of pain in the test stimulus.The conditioned pain modulation will be performed at two different times: before and after the single tDCS onset.
Change in the quantitative sensory test (QST) | Up to 60 minutes after tDCS onset.
  The quantitative sensory test (QST) evaluates the function of myelinated, small and unmyelinated fibers, also including the function of the spinothalamic tract and nociceptive fibers. In addition, the QST represents a non-invasive method, which determines the gain or loss of sensory perception in response to external stimuli of controlled intensity in a previously determined body area.
  The following tests will be carried out in the research:
  * Painful pressure threshold: performed with a pressure algometer, applied on the upper extremity.
  * Cold pressor test: the patient puts his extremity in a container with ice. The tolerance time will be determined.
  * Sensation of heat: using a heat electrode applied to the extremity corresponding to the sensitive alteration, the first sensation of heat and the painful threshold of light, medium and maximum heat will be evaluated.
  The QST measures will be performed at two different times; before and after the tDCS onset.

OTHER OUTCOMES:
levels of Brain derived neurotrophic factor | Blood samples will be collected at baseline, before tDCS onset.
  Blood samples will be collected at baseline in order to determine BDNF serum levels using a standardized kit

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bishop JM, Levinson WE, Quintrell N, Sullivan D, Fanshier L, Jackson J. The low molecular weight RNAs of Rous sarcoma virus. I. The 4 S RNA. Virology. 1970 Sep;42(1):182-95. doi: 10.1016/0042-6822(70)90251-5. No abstract available. PMID 4318979
- [Background] van Dun K, Bodranghien FC, Marien P, Manto MU. tDCS of the Cerebellum: Where Do We Stand in 2016? Technical Issues and Critical Review of the Literature. Front Hum Neurosci. 2016 May 11;10:199. doi: 10.3389/fnhum.2016.00199. eCollection 2016. PMID 27242469
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Background] Lefaucheur JP. Transcranial magnetic stimulation. Handb Clin Neurol. 2019;160:559-580. doi: 10.1016/B978-0-444-64032-1.00037-0. PMID 31277876
- [Background] Ugawa Y, Day BL, Rothwell JC, Thompson PD, Merton PA, Marsden CD. Modulation of motor cortical excitability by electrical stimulation over the cerebellum in man. J Physiol. 1991 Sep;441:57-72. doi: 10.1113/jphysiol.1991.sp018738. PMID 1816387
- [Derived] Betancur DFA, da Graca Lopes Tarrago M, Franca BR, Bueno GB, Gomes J, Coelho ML, Venturini CL, Torres ILS, Fregni F, Bock H, Caumo W. Cortical excitability and analgesic effects of multisite transcranial direct current stimulation targeting the motor cortex and cerebellum in fibromyalgia. Sci Rep. 2025 Oct 23;15(1):37067. doi: 10.1038/s41598-025-20769-1. PMID 41130992